CLINICAL TRIAL: NCT02494726
Title: Prospective Analysis of the Use of Thromboelastography in Stroke Patients
Brief Title: Prospective Analysis of the Use of TEG in Stroke Patients
Acronym: TEG
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James Grotta, Professor and Chair, Department of Neurology, The University of Texas Health Science Center, Houston
Other Study IDs: MS-09-0156
Record Dates: First submitted 2015-07-04; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Stroke; Brain Hemorrhage
Keywords: Ischemic stroke; ICH stroke; TEG; Thromboelastography; Stroke
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages; Stroke | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ischemic Stroke: Ischemic stroke patients who have had blood analyzed using thromboelastography (TEG)
  Interventions: Other: Thromboelastography
- Healthy Controls: Healthy controls who have had their blood analyzed using thromboelastography (TEG)
  Interventions: Other: Thromboelastography
- Hemorrhagic Stroke: Intracerebral hemorrhage patients who have had their blood analyzed by thromboelastography (TEG)
  Interventions: Other: Thromboelastography

INTERVENTIONS:
Other: Thromboelastography — TEG (Thrombelastography) measurements include: Split Point (SP) is the time elapsed for the clot to initially form fibrin when the blood is first placed in the TEG machine. Reaction Time (R) is the time elapsed from its initial fibrin formation until the clot reaches 2mm. K is the time measured from R until the level of clot firmness reaches 20mm, measuring the speed of clot strengthening. These are measured in minutes. Delta measures if the formation of the clot has been suppressed; measured as the difference between R and SP. Angle reflects the speed at which clots form by forming the slope of the TEG tracing at R from the horizontal line. Maximum Amplitude (MA) in mm is the measure of maximum strength of the clot, true platelet function. G is the measure of the clot firmness; measured by a formula (G=(5000*MA)/(100-MA) in dynes/cm2). LY30 is a measure of clot lysis at 30 minutes after MA is reached.
  Other Names: TEG

SUMMARY:
The overall purpose of this study is to evaluate how effective Thromboelastography (TEG) is on identifying ischemic and hemorrhagic stroke patients at increased risk for bleeding after receiving tissue plasminogen activator (tPA), as well as on differentiating between patients in whom optimal thrombolysis has been achieved, and those whom it has not.

DETAILED DESCRIPTION:
Thromboelastography (TEG), a computerized analysis that has been used since the 1940s, is the only stand alone test that can provide integrated information on the balance between the two separate but simultaneously occuring components of coagulation, thrombosis and lysis. It measures the coagulation process from initial clotting cascade to clot strength.

TEG may be used to assess the coagulation status of patients with acute stroke, whether ischemic or hemorrhagic. TEG might also be a useful way to predict and assess the degree of fibrinolysis that is achieved by tissue plasminogen activator (tPA). Currently tPA is given as a standard dose determined by the patient's body weight, thus given the variability in patient outcome after tPA, this dose could sometimes be too small or too large, leading to thrombolysis or bleeding, respectively. One of the purposes of this observational study is to evaluate how effective TEG is on predicting and assessing the degree of thrombolysis following tPA therapy, by producing a range of TEG values correlated with optimal thrombolysis.

The results of the recent FAST trial demonstrated the need to identify patients with spontaneous intracerebral hemorrhage (ICH) who are at increased risk for hematoma enlargement. Such identified patients, could benefit from a therapeutic advantage of activated factor VII or other hemostatic agents may be more clearly studied. Therefore, another purpose of this study is to evaluate how effective TEG is on predicting further bleeding for patients with spontaneous ICH.

The study will consist of 208 ischemic patients and 80 hemorrhagic patients, whom which are approached from all stroke patients admitted to Memorial Hermann Hospital Emergency Department receiving a confirmatory CT or MRI scan. Patients who agree to participate will have blood drawn the day of hospital arrival, will then be followed for 36 +/- 12 hours after the stroke, and 90 +/- 30 days after the stroke, all during which two more blood samples will be obtained.

Normal controls will be age and sex matched to the investigators' research population. A one-time blood draw will be obtained and information collected will be age, sex and TEG values.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older.
* Symptoms and signs causing measurable neurologic deficit consistent with an acute stroke.
* CT or MRI consistent with stroke (ischemic or hemorrhagic) or with clinical evidence suggesting a stroke.
* For acute ischemic stroke patients, treatment with tPA and TEG blood draw must be done within 4.5 hours of symptom onset.
* For ICH patients, TEG blood draw must be done within 6 hours of symptom onset.

Exclusion Criteria:

* Contraindication to CT and MRI (ex. inability to lie flat)
* If ICH patient
* Hemorrhage secondary to trauma, arteriovenous malformation (AVM) or crush injury
* Planned surgical evacuation (hemicraniectomy and ventriculostomy allowed).
* Receipt of hemostatic agents (FFP, Cryo, activated factor seven) prior to TEG blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All stroke patients admitted to Memorial Hermann Hospital Emergency Department receiving a confirmatory CT or MRI scan.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2009-11; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Baseline TEG in patients with spontaneous ICH vs age matched controls | TEG obtained within 6 hours of last seen normal in patients with spontaneous ICH
  Compare baseline (within 6 hours of last seen normal) TEG in patients with spontaneous ICH to TEG in age-matched controls.

SECONDARY OUTCOMES:
Rapid clinical improvement after tPA (8 or greater point improvement on NIHSS score or total NIHSS 0 or 1) | Change in NIHSS score from baseline (prior to IV tPA within 4.5 hours of last seen normal) to NIHSS 36 +/- 12 hours after last seen normal.
  Correlate baseline (within 4.5 hours of last seen normal and prior to tPA) and 10 minute post tPA TEG values with rapid clinical improvement

OTHER OUTCOMES:
Hematoma enlargement in patients with spontaneous ICH | CT hematoma volume at 36 +/- 12 hours compared to baseline (within 6 hours of last seen normal)
  Correlate baseline TEG values (within 6 hours of last seen normal) with hematoma enlargement
Hemorrhagic transformation after IV tPA | Any bleeding on post tPA imaging 36 hours +/- 12 hrs after stroke onset
  Correlate baseline TEG values (within 4.5 hours of last seen normal) with hemorrhagic transformation or hemorrhage on CT 36 hours after stroke onset
Arterial recanalization after IV tPA | Recanalization (TICI 2b or 3 flow) on imaging within 36 hours post IV tPA compared to pre-treatment
  Correlate baseline TEG values (within 4.5 hours of last seen normal) with recanalization (TICI 2b or 3 flow) on imaging within 36 hours post IV tPA compared to pre-treatment
Hyperdense Middle Cerebral Artery Sign (HDMCA) | HDMCA on baseline CT in patients receiving IV tPA within 4.5 hours of last seen normal
  Correlate baseline TEG values (within 4.5 hours of last seen normal) with HDMCA on baseline CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: James Grotta, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Medical School at Houston, Houston, Texas, United States